CLINICAL TRIAL: NCT01232712
Title: A Novel Vaccine for the Treatment of MUC1-expressing Tumor Malignancies
Brief Title: A Study to Assess the Safety and Efficacy of MUC1 Peptide Vaccine and hGM-CSF in Patients With MUC1-positive Tumor Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaxil Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAXIL-001
Record Dates: First submitted 2010-10-22; First posted 2010-11-02 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Myeloma
Keywords: MUC1; ImMucin; Vaccine; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ImMucin (Experimental): Treatment with ImMucin and rhGMCSF (recombinant human granulocyte-monocyte colony stimulating factor)
  Interventions: Biological: ImMucin, hGM-CSF

INTERVENTIONS:
Biological: ImMucin, hGM-CSF — * Six biweekly Intradermal or subcutaneous injections of 100 micrograms ImMucin
  * After six injections, if response will not be observed, or if response will not be sufficient, Immucin dose will be escalated to 250 micrograms for six additional injections.
  * In addition, each immunization, hGM-CSF with a total dose of 250 microgram will be injected.

SUMMARY:
The scientific approach behind this study is to develop novel anti-cancer therapeutic vaccine to induce a robust cellular immune response mediated via both CD4+ and CD8+ T lymphocytes populations and can be be applicable to the majority of the target population.

ELIGIBILITY:
Inclusion Criteria:

1. All* patients must have a histological or cytological diagnosis of metastatic disease or hematological malignancies expressing the MUC1. Patients must have metastatic disease, and have failed at least one regimen of standard based chemotherapy for metastatic disease as indicated in the following table. Patients must have disease considered to be incurable by surgical or radiological intervention.
2. Patients must be > 18 years of age, consenting to participate in the study.
3. Patients must have at least one site of measurable tumor or measurable tumor marker.
4. Radiological and other relevant imaging studies, such as CT scans, must be performed within 4 weeks of the first treatment as a baseline to document extent of disease.
5. Patients should be at least 4 weeks beyond any major surgery or chemoradiotherapy and have recovered from drug induced toxicity.
6. Patients must have a performance status of 70% or greater on the Karnofsky scale (ECOG 0-2) and a minimal life expectancy of 12 months.
7. Patients must sign an informed consent, and be mentally responsible.

   * In Multiple Myeloma, MUC1 expression will be tested after confirming that all inclusion/exclusion criteria are met and within the screening period.

Exclusion Criteria:

1. Patients not fulfilling the above criteria.
2. Patients with a significant concurrent medical complication that in the judgment of the Principal Investigator could affect the patient's ability to tolerate or complete this study.
3. Patients receiving any immunosuppressive treatment that could negate development of an effective immune response to the vaccine. (First vaccination should be at least 30 days from end of immunosuppressive treatment)
4. Subjects with prior irradiation to a field that includes more than 25% of their lymph nodes and bone marrow likely to be immunosuppressed will be excluded. However, patients who had standard pelvic field radiation as adjuvant therapy for rectal cancer are not excluded.
5. Pregnant and breast feeding women will be excluded. Premenopausal women who are not practicing or willing to practice adequate birth control methods for a period of 3 months after treatment will be excluded.
6. Patients with brain metastasis.
7. Patients with active infection.
8. Patients with HIV HBSAg and HCV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety of intradermal or subcutaneous administration of the ImMucin peptide | 6 months
  Determine the safety and initial feasibility of intradermal or subcutaneous administration of the ImMucin peptide combined with hGM-CSF for maximal stimulation of T cell response.
  The patients will receive six or twelve biweekly injections of Imucin (3 or 6 months). Post Treatment visit will be performed 4 weeks after administration of last vaccination. FU telephone calls will be made up to 6 months following the last vaccination in order to assess the status of the disease.

SECONDARY OUTCOMES:
Assess efficacy of study treatment | 6 months
  Assessment of respose to treatment during treatment period (3 or 6 months).Post Treatment visit will be performed 4 weeks after administration of last vaccination. FU telephone calls will be made up to 6 months following the last vaccination in order to assess the status of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

REFERENCES:
- See also: Vaxil BioTherapeutics Ltd. web site — http://www.vaxilbio.com